CLINICAL TRIAL: NCT01272453
Title: Computed Tomography Dose Reduction Using Sequential or Fast Pitch Sprial Technique Employed in Cardiothoracic Imaging
Brief Title: Computed Tomography Dose Reduction Using Sequential or Fast Pitch Sprial Technique
Acronym: CTDOSE
Status: Completed | Type: Observational
Sponsor: Gilbert L. Raff, MD (Other)
Collaborators: Siemens Healthcare Diagnostics Inc (Industry)
Responsible Party: Sponsor-Investigator, Gilbert L. Raff, MD, Medical Director, Advanced Cardiovascular Imaging, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2010-209
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease; Aortic Aneurysm; Pulmonary Embolism
Keywords: coronary artery disease; CT scan; coronary angiography; chest pain; aortic aneurysm; pulmonary embolism
MeSH Terms: conditions — Coronary Artery Disease; Aortic Aneurysm; Pulmonary Embolism; Chest Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Data from patients in the control group will be obtained retrospectively from patient medical records and stored image data
- Prospective Patient Group: Data from patients in the Flash group will be obtained prospectively from scanner consoles and medical records.

SUMMARY:
This is a prospective, controlled observational trial of patients undergoing clinically indicated cardiothoracic computed tomography (CT), including pulmonary or aortic angiography and coronary CT angiography (CCTA).

DETAILED DESCRIPTION:
The development of a novel CT scanner capable of sequential or fast-pitch spiral techniques in most patients (Siemens Definition Flash) represents a potentially crucial technical innovation at a particularly critical juncture. National healthcare systems are under pressure to deliver accurate and cost-effective diagnosis of an increasing number of patients and CT angiography in various settings is a proven, highly accurate technique that has been shown to improve diagnostic efficiency and reduce the cost of care.

However, there has been increasing concern about the lifetime attributable risk of cancer from radiation related to diagnostic procedures. Such concern extends to other radiation-based procedures that contribute to the cumulative lifetime radiation exposure of patients. The Flash scanner holds the promise of substantially reducing exposure resulting from a variety of examinations.

The CT DOSE multicenter trial is therefore designed to validate the extent of dose reduction attendant to the use of the Flash scanner in cardiothoracic scanning, and to determine whether image quality is preserved in spite of significant dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* Scans from patients undergoing clinically indicated pulmonary angiography, aortography and/or CCTA.
* Age greater than or equal to 18 years.

Exclusion Criteria:

* No exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically indicated cardiothoracic computed tomography (CT), including pulmonary or aortic angiography and coronary CT angiography (CCTA)at 10 sites. Patient selection will be based on a site consecutive CT scan log.
Sampling Method: Non-Probability Sample
Enrollment: 2640 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Radiation dose | Time of CT scan
  The primary endpoint is radiation dose, measured as dose-length-product (DLP, in mGy∙cm) and effective radiation dose, calculated as DLP x 0.014 (in mSv).

SECONDARY OUTCOMES:
Assessment of Image Quality | Time of CT Scan
  Signal noise (standard deviation of attenuation in Hounsfield units) will be determined in regions of interest in: A) air anterior to the chest wall, B) mid-LV septum and C) mid thoracic aorta or main PA. This will be done in a sequential sample of every 5th case (approximately 600 cases total).

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Raff, MD, Principal Investigator — Corewell Health East
Locations (9):
- United States (8):
  - Naval Medical Center, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Troy, Troy, Michigan
  - Minneapolis Heart Institute/ Abbott Northwestern, Minneapolis, Minnesota
  - NYU Langone Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
- King Abdul-Aziz Cardiac Center, national Guard Health Affairs, Riyadh, Kingdom of Saudi Arabia, Saudi Arabia